CLINICAL TRIAL: NCT04376775
Title: Assessment of the Impact of COVID-19 on Transplant Patients and on Patients Awaiting Transplantation
Acronym: COWAIT
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Société Francophone de Transplantation (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/19
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Transplantation
Keywords: Waiting list; Transplantation; Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transplant patient: This study will involve all the transplant centres in France. The investigator will use patient-completed surveys for all participants. Wait Listed Transplant Candidates and Transplant Recipients (liver, kidney, pancreas, heart, lung) will be contacted by the all French transplant centres and patient's associations.
  Interventions: Other: Transplant patient

INTERVENTIONS:
Other: Transplant patient — Surveys will be distributed via an email sent by transplant centres or patient's associations. A link to a secure survey platform will be given. A questionnaire will completed by patients. Patients, who agreed to fill the survey, will be offered the possibility to be contacted for a second survey over a 6 months period.

SUMMARY:
To provide optimal care to patients and to maintain long-term institutional viability, Transplant Centres (TC) must have an awareness of their patients' health status, their health care needs and priorities, as well as their access to information and health care. For example, it is critical that TCs understand whether their patients are medically suitable for transplant, whether transplantation remains a priority for their patients, how best to communicate with their patients, and whether their patients have sufficient access to medications and health care to undergo transplant safely. The COVID-19 pandemic has had a tremendous impact on people and institutions around the country in a short period of time. At this time, little is known regarding its impact on the transplant community specifically. For example, it has been reported that around 8 million French applied for partial unemployment benefit over the past month, but it is not known if this has affected transplant patients. It has been reported that people with significant chronic medical conditions and those with compromised immune systems may be at increased risk of dying from the COVID-19, but it is not known if this has affected patients' interest in receiving transplants at this time. The "Société Francophone de Transplantation (SFT)" published recommendations at the beginning of the pandemic in order to limit the rate of infection in these high-risk population. The purpose of this study is to better understand the impact of COVID-19 on patients on the waiting list and transplant patients. Further, a better understand on how patients have received information about this pandemic and how best to communicate with them.

DETAILED DESCRIPTION:
Transplant Centres (TCs) serve a unique patient population, those with end-organ disease who are either waiting for, or who have received, a solid-organ transplant. For transplant candidates, TCs help weigh the threat of their current condition against the intended benefits and associated risks of transplantation, which include major-surgery and chronic immune suppression (IS). For transplant recipients, TCs help manage the life-long risks associated with IS, including infection and malignancy, and facilitate access to appropriate health care over time.

To provide optimal care to patients and to maintain long-term institutional viability, TCs must have an awareness of their patients' health status, their health care needs and priorities, as well as their access to information and health care. For example, it is critical that TCs understand whether their patients are medically suitable for transplant, whether transplantation remains a priority for their patients, how best to communicate with their patients, and whether their patients have sufficient access to medications and health care to undergo transplant safely.

The COVID-19 pandemic has had a tremendous impact on people and institutions around the country in a short period of time. At this time, little is known regarding its impact on the transplant community specifically. For example, it has been reported that around 8 million French applied for partial unemployment benefit over the past month, but it is not known if this has affected transplant patients. It has been reported that people with significant chronic medical conditions and those with compromised immune systems may be at increased risk of dying from the COVID-19, but it is not known if this has affected patients' interest in receiving transplants at this time. The "Société Francophone de Transplantation (SFT)" published recommendations at the beginning of the pandemic in order to limit the rate of infection in these high-risk population. Briefly, these recommendations encompassed the following points: Not stopping immunosuppression, strict application of the social distancing, recommendation to stay and work at home, recommendation to limit the visits at the hospital. However, it is still unclear whether these recommendations were followed by the transplant recipients, and if this exceptional situation has affected their access to health care or needed medications.

The purpose of our study is to better understand the impact of COVID-19 on patients on the waiting list and transplant patients. Further, a better understand on how patients are receiving information about this pandemic and how best to communicate with them. The hypothesis is that peri-transplant patient groups may appropriately perceive themselves to be at high risk of infection and poor outcomes, and that this may influence their decisions around seeking medical care and willingness to undergo organ transplantation. Additionally, the investigator anticipate a wide range of needs and risks among patients, including their ability to isolate from potential infection, ability to access medications and medical care, and their ability to access information regarding COVID-19. Ultimately, the investigator plan to use the information collected from patients to improve patient education regarding COVID-19 and to inform centres' response to future epidemics and/or natural disasters that disrupt patient care. Until now, no systematic description of transplant patients' needs, priorities, behavior's, attitudes, or education has been done during this pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Patients currently (at the time of survey) on a French transplant waiting list.
* Patients transplanted with a functional graft.

Exclusion Criteria:

* Under 18 years of age,
* Patients under protective measures or deprived of their liberty:

pregnant or breastfeeding woman, under guardianship, under curatorship, safeguard of justice, incarcerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients registered on the French waiting list for a transplant and patients transplanted with a functional graft.
Sampling Method: Non-Probability Sample
Enrollment: 3602 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Compliance precautions with COVID-19 | In a maximum of 6 months after inclusion
  The compliance will be assessed by the questionnaire created for the study. The questionnaire has 38 questions with multiple choice for each question.

SECONDARY OUTCOMES:
Clinical impact of COVID-19 | In a maximum of 6 months after inclusion
  The clinical impact will be assessed by the questionnaire created for the study. The questionnaire has 38 questions with multiple choice for each question.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pellegrin, Bordeaux, France